CLINICAL TRIAL: NCT05244772
Title: Quality of Recovery After Day Care Surgery With App Controlled Remote Monitoring: a Randomized Controlled Trial
Acronym: QuReMo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Responsible Party: Principal Investigator, M.B. Godfried, Anesthesiologist, Onze Lieve Vrouwe Gasthuis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL78144.100.21 / WO21.083
Record Dates: First submitted 2022-02-09; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Pain; Nausea; Vomiting
Keywords: eHealth; Remote monitoring; Anaesthesia; Day care surgery
MeSH Terms: conditions — Pain; Nausea; Vomiting | interventions — Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote monitoring (Experimental): At discharge, patients in the remote monitoring group receive verbal and paper care- and recovery instructions from a day care ward nurse and in adittion they will have a monitoring application installed on theirpersonal smartphone. Once they are back home, they can start recording pain and nausea and ask questions about their recovery with the application and report back the anaesthesia backoffice.
  Interventions: Other: Remote monitoring
- Standard care (No Intervention): At discharge, patients in the standard care group receive verbal and paper care- and recovery instructions from a day care ward nurse.

INTERVENTIONS:
Other: Remote monitoring — Remote monitoring with a smartphone application of pain and nausea after day care surgery
  Arms: Remote monitoring

SUMMARY:
Non blinded randomized controlled trial with mixed methods design. To assess the experienced quality of recovery after day care surgery between patients provided with remote home monitoring and patients receiving standard discharge care

DETAILED DESCRIPTION:
Rationale: To date the majority of surgical interventions is performed in day care and patients are being discharged soon after the first critical postoperative period. At home, patients have limited options to contact the hospital in case of severe pain and nausea. We have provided day care surgical patients with a smartphone application for remote monitoring that is configured to self-record postoperative pain and nausea after being discharged from hospital. Furthermore, it provides a messaging service to contact the hospital in case of (severe) pain or nausea. Despite the promising initial patient experiences of such an application, we do not know whether remote monitoring with a smartphone application improves the patient's experience during the recovery period.

Objective: To evaluate the experienced quality of recovery after day care surgery between patients provided with a smartphone application for remote monitoring and patients receiving standard of care (no remote monitoring).

Study design: (Non-blinded) randomized controlled trial with mixed methods design Study population: Adult patients (aged 18 years or older) scheduled for day care surgery Intervention (if applicable): The intervention group receives the smartphone application for remote monitoring during weekdays from 8 am to 17 pm up to 7 days after surgery. With this application, patients are able to record experienced pain and nausea. In addition, they can send messages to the hospital. Daily monitoring is performed by an anaesthesia professional who will contact the patient in case severe pain or nausea is reported in the app. The control group receives standard of care (with post-discharge verbal and paper instructions).

Main study parameters/endpoints: The main study endpoint is the difference between patients using remote monitoring and patients not using remote monitoring in perceived quality of recovery measured with the QoR-15 questionnaire on the 7th day after day care surgery. Secondary endpoints are 1) the overall score on the Quality of Recovery-15 at day 1, 4 and 7 post discharge, 2) the perceived quality of hospital aftercare and 3) experienced psychological effects of remote monitoring during postoperative recovery from day care surgery.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participating in this study does not pose any additional risks either for patients allocated to the intervention group with remote monitoring or for patients allocated tothe standard of care group. Patients in the remote monitoring group are being asked to use a smartphone application to record pain and nausea daily for up to 7 days post discharge. Recording pain and nausea will take 2 minutes daily. Patients from both groups are being asked to fill in the validated QoR-15 questionnaire one day before admission and on the 1st, 4th and 7th day post discharge and this will take 2.5 minutes. No extra hospital visits, physical examinations or tests are required. Patients in the remote monitoring group could benefit from participating in the study because they are monitored daily by a healthcare professional. Therefore, severe pain, nausea and possibly other complications can be noticed and managed earlier.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Age: older than or equal to 18 years
* Pre-anaesthesia conclusion: ASA I to III
* Scheduled for day care surgery for one of the following surgical specialties:

gynaecology, eye-nose and throat, oral and maxillofacial, orthopaedics, general and vascular, trauma and urology -In possession of a smartphone

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Not able to speak or understand the Dutch language
* Mentally impaired (e.g. dementia, retardation)

During study:

-Patients who experience a unexpected post-operative complication or prolonged recovery with the result that discharge on the same day of the surgical intervention is not possible will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery | 7th day after day care surgery
  To assess the difference between patients using remote monitoring and patients not using remote monitoring in perceived quality of recovery measured with the QoR-15 questionnaire on the 7th day after day care surgey

SECONDARY OUTCOMES:
Postoperative pain | 1st, 4th and 7th day after day care surgery
  To assess the experienced postoperative pain (POP) between patients provided with a smartphone application for remote monitoring and patients receiving standard of care (no remote monitoring) after day care surgery.
Post discharge nausea and vomiting | 1st, 4th and 7th day after day care surgey
  To assess the experienced post discharge nausea and vomiting (PDNV) between patients provided with a smartphone application for remote monitoring and patients receiving standard of care (no remote monitoring) after day care surgery.
Surgical complications | 1st 4th and 7th day after day care surgey
  To assess the difference in the number of surgical complications rated with the Clavien Dindo classification of surgical complication between patients provided with a smartphone application for remote monitoring and patients receiving standard of care (no remote monitoring) after day care surgery.
Re-admissions | 1st, 4th and 7th day after day care surgery
  To assess the difference in the number of re-admissions between patients provided with a smartphone application for remote monitoring and patients receiving standard of care (no remote monitoring) after day care surgery.
Contact with healthcare professionals | 1st, 4th and 7th day after day care surgey
  To assess the difference in the number of hospital contacts / general practitioner between patients provided with a smartphone application for remote monitoring and patients receiving standard of care (no remote monitoring) after day care surgery.
Experienced communication | 1st, 4th and 7th day after day care surgey
  To assess the difference in experienced quality of communication with the hospital staff between patients provided with a smartphone application for remote monitoring and patients receiving standard of care (no remote monitoring) after day care surgery.
Experienced psychological effects | 1st, 4th and 7th day after day care surgey
  o assess the experienced psychological effects remote monitoring in patients recovering from day care surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Godfried, PhD, Principal Investigator — OLVG Hospital; Seppe Koopman, PhD, Principal Investigator — Maasstad Hospital; Robert van Dongen, PhD, Principal Investigator — CWZ Hospital
Locations (3):
- Netherlands (3):
  - CWZ Hospital, Nijmegen, Limburg
  - OLVG Hospital, Amsterdam, North Holland
  - Maasstad Hospital, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Yes
The study will be registered before inclusion of the first patient on www.clinicaltrials.gov. The results of the study will find their way into (inter-) national scientific journals and guidelines. We will submit analyses to scientific journals in the field of anaesthesiology.
Supporting Information: Study Protocol, CSR
Time Frame: Available december 2022
Access Criteria: Request for information can be adressed to b.thiel@olvg.nl.

REFERENCES:
- [Derived] Thiel B, Godfried M, van Emst M, Vernooij L, van Vliet L, Rumke E, Snoeck M, Koopman S, Kalkman C. Discharge with a smartphone application for follow-up after day care surgery: a randomised controlled trial. BJA Open. 2025 Sep 25;16:100489. doi: 10.1016/j.bjao.2025.100489. eCollection 2025 Dec. PMID 41079519
- [Derived] Thiel B, Godfried MB, van Emst ME, Vernooij LM, van Vliet LM, Rumke E, van Dongen RTM, Gerrits W, Koopman JSHA, Kalkman CJ. Quality of recovery after day care surgery with app-controlled remote monitoring: study protocol for a randomized controlled trial. Trials. 2023 Feb 9;24(1):102. doi: 10.1186/s13063-023-07121-6. PMID 36759858

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT05244772/Prot_SAP_000.pdf